CLINICAL TRIAL: NCT01898234
Title: Assessment of Subjective and Hemodynamic Tolerance of Different High- and Low-flux Dialysis Membranes in Patients Undergoing Chronic Intermittent Hemodialysis: a Randomized Controlled Trial
Brief Title: Dialysis Membranes and Hemodynamic Tolerance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale Regionale di Locarno (Other)
Responsible Party: Principal Investigator, Luca Gabutti, MD, Prof, Head of Department of Internal Medicine, Ospedale Regionale di Locarno
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 012012
Record Dates: First submitted 2013-07-02; First posted 2013-07-12 (Estimated); Last update posted 2013-07-12 (Estimated); Status verified 2013-07

CONDITIONS: Dialysis Membranes and Hemodynamic Tolerance
Keywords: Hemodynamics; intradialytic hypotension; subjective tolerance; dialysis membranes; high flux; low flux; hemodialysis

ARMS (4):
- Revaclear (Experimental)
  Interventions: Device: Revaclear
- Helixone high flux (Experimental)
  Interventions: Device: Helixone high flux
- Xevonta (Experimental)
  Interventions: Device: Xevonta
- Helixone low flux (Experimental)
  Interventions: Device: Helixone low flux

INTERVENTIONS:
Device: Revaclear — Four polysulfone dialyzers of 1.8 m2, A (Revaclear, Gambro), B (Helixone high flux, Fresenius), C (Xevonta, BBraun) and D (Helixone low flux, Fresenius), were compared with each other
  Other Names: -Revaclear, Gambro 1.8 m2
  Arms: Revaclear
Device: Helixone high flux — Four polysulfone dialyzers of 1.8 m2, A (Revaclear, Gambro), B (Helixone high flux, Fresenius), C (Xevonta, BBraun) and D (Helixone low flux, Fresenius), were compared with each other
  Other Names: Helixone high flux, Fresenius 1.8 m2
  Arms: Helixone high flux
Device: Xevonta — Four polysulfone dialyzers of 1.8 m2, A (Revaclear, Gambro), B (Helixone high flux, Fresenius), C (Xevonta, BBraun) and D (Helixone low flux, Fresenius), were compared with each other
  Other Names: Xevonta, BBraun 1.8 m2
  Arms: Xevonta
Device: Helixone low flux — Four polysulfone dialyzers of 1.8 m2, A (Revaclear, Gambro), B (Helixone high flux, Fresenius), C (Xevonta, BBraun) and D (Helixone low flux, Fresenius), were compared with each other
  Other Names: Helixone low flux, Fresenius 1.8 m2
  Arms: Helixone low flux

SUMMARY:
Background:

High- and low-flux dialysis membranes made of different materials may correlate with various hemodynamic tolerance profiles. This study aims to investigate hemodynamic response and incidence of hypotensive episodes by comparing some of the most commonly used high- and low-flux dialyzers.

Methodology:

The study was designed as an open label, randomized, cross-over investigation, including 25 patients undergoing chronic hemodialysis. Four polysulfone dialyzers of 1.8 m2, A (Revaclear, Gambro), B (Helixone high flux, Fresenius), C (Xevonta, BBraun) and D (Helixone low flux, Fresenius), were compared with each other. The hemodynamic profile was assessed with a non-invasive technique and patients were asked to provide tolerance feedback through a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* age 18 and older
* ability to understand the information presented and sign the informed consent
* chronic hemodialysis for at least 8 weeks
* stable dialysis prescriptions and modality in the 2 weeks prior to protocol implementation

Exclusion Criteria:

* mental illness;
* inability to understand the information presented and sign the informed consent;
* acute disease requiring hospitalization at the time of patient enrolment
* pregnancy and breast feeding

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-10; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
comparative evaluation of mean hemodynamic parameters (i.e. systolic and diastolic blood pressure, peripheral resistance and cardiac output) during dialysis | 4 weeks
comparative evaluation of subjective tolerance across the various membranes | 4 weeks
  As to the assessment of subjective tolerance, we decided to administer the questionnaire designed by Cruz et al. [Cruz DN, Mahnensmith RL, Brickel HM, Perazella MA. Midodrine and cool dialysate are effective therapies for symptomatic intradialytic hypotension. Am. J. Kidney Dis. 1999 Mag;33(5):920-926] then modified by Teruel et al. [Teruel JL, Martins J, Merino JL, Fernández Lucas M, Rivera M, Marcén R, et al. Temperature of the dialysis bath and hemodialysis tolerance. Nefrología: PublicaciónOficial De La Sociedad Española Nefrologia. 2006;26(4):461-468] and to integrate it with a 1 to 10 numerical scale to assess patient well-being
comparative evaluation of Kt/V and of beta-2 microglobulin removal | 4 weeks

SECONDARY OUTCOMES:
comparative analysis of the incidence of symptomatic and non-symptomatic systolic pressure drops (> 20 mmHg) | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Luca Gabutti, MD, Principal Investigator — Ospedale Regionale Locarno
Locations (1):
- Ospedale Regionale di Locarno, Locarno, Canton Ticino, Switzerland